CLINICAL TRIAL: NCT04987463
Title: Randomized, Placebo-controlled, Double-blind and Double-dummy Clinical Trial Comparing the Safety, Tolerability, and Efficacy of Vigabatrin and Rapamycin in a Preventive Treatment of Infants With Tuberous Sclerosis Complex
Brief Title: Efficacy and Safety of Rapamycin Versus Vigabatrin in the Prevention of Tuberous Sclerosis Complex Symptoms in Infants
Acronym: ViRap
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Katarzyna Kotulska (Other)
Responsible Party: Sponsor-Investigator, Katarzyna Kotulska, Head of the Department of Neurology and Epileptology at The Children's Memorial Health Institute, Children's Memorial Health Institute, Poland
Organization: Children's Memorial Health Institute, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ViRap
Record Dates: First submitted 2021-05-28; First posted 2021-08-03 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Tuberous Sclerosis Complex
Keywords: tuberous sclerosis complex, epilepsy, rapamycin, vigabatrin, tumors, prevention
MeSH Terms: conditions — Tuberous Sclerosis; Epilepsy; Neoplasms | interventions — Vigabatrin; Sirolimus; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vigabatrin arm (Experimental): Vigabatrin in capsules co-administered with placebo in liquid.
  Interventions: Drug: Vigabatrin; Drug: Placebo
- Rapamycin arm (Experimental): Rapamycin in liquid co-administered with placebo in capsules.
  Interventions: Drug: Rapamycin; Drug: Placebo

INTERVENTIONS:
Drug: Vigabatrin — Vigabatrin in capsules administered orally, initially (between V1 and V2) once daily in the evening,and starting from V2 administered two times daily.
  Arms: Vigabatrin arm
Drug: Rapamycin — Rapamycin in liquid administered orally, in the morning, every other day or daily depending on the patient's body weight. The starting dose of rapamycin will be calculated according to the body weight of the patient measured at V1.
  Arms: Rapamycin arm
Drug: Placebo — Placebo in liquid administered orally, once daily, in the morning. The starting dose of placebo in liquid will be calculated according to the body weight of the patient measured at V1.
  Other Names: Placebo in liquid
  Arms: Vigabatrin arm
Drug: Placebo — Placebo in granules administered orally, initially once daily in the evening,and after reaching the targeted dose administered two times daily.
  Other Names: Placebo in granules
  Arms: Rapamycin arm

SUMMARY:
The purpose of the study is to evaluate the efficacy, tolerability, and safety of vigabatrin versus rapamycin as a preventive treatment in infants with Tuberous Sclerosis Complex (TSC).

DETAILED DESCRIPTION:
This is a two-arm, randomized, double-blind and double-dummy, placebo controlled study to evaluate the efficacy, tolerability, and safety of vigabatrin versus rapamycin as a preventive treatment in infants with TSC. The study consists of 3 phases for each patient: screening, core blinded phase, and open-label follow-up phase. Patients who meet the eligibility criteria will be randomized to receive vigabatrin or rapamycin. The randomization ratio is 1:1. Randomization will be stratified by the sex and the presence of epileptiform activity on baseline videoEEG (video electroencephalography) recording (yes versus no). Approximately 60 infants are planned to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 4 up to 16 weeks (44-56 weeks of gestational age) at the day of randomization
* Parents/caregivers are willing to and able to give informed consent form for the participation in the study
* Parents/caregivers are willing to and able to comply with all study requirements
* Definite diagnosis of TSC according to the Consensus criteria (Northrup,2013)
* At least 1 focus of cortical dysplasia disclosed on brain MRI

Exclusion Criteria:

* history of seizures prior to randomization,
* history of antiepileptic treatment,
* history of treatment with mTOR (mammalian Target of Rapamycin) inhibitor,
* gestational age below 44 weeks at the day of randomization,
* body weight lower than 3 kg at the day of randomization,
* SEGA (Subependymal Giant Cell Astrocytoma) or other TSC-associated lesion requiring urgent surgical intervention
* recent surgery within 1 month prior to the randomization
* intercurrent infection at the date of randomization
* known history of HIV seropositivity
* live vaccination within 1 month prior to randomization*
* lack of first TBC and hepatitis B vaccinations
* Any significant clinical, laboratory , ECG or other abnormalities, comorbidity or concomitant treatment which, in the opinion of the investigator, may either put a patient at significant risk associated with the participation in the study or may influence the results of the study.
* Use of an investigational drug within 1 month prior to randomization.

Ages: 4 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of clinical seizures in the blinded phase of the study, | 730 days
Summarized volume of TSC-associated tumors ≥ 125% of initial value within the blinded phase of the study | 730 days

SECONDARY OUTCOMES:
Total volume of TSC-associated tumors within the blinded phase and the whole study | 730 days
The risk for high risk of autism assessed with psychological test at 6, 12, 18, 24 months | 6, 12, 18, 24 months
The risk for low developmental quotient (< 70 points in Bayley Scales of Infant Development, measured at the end of the blinded phase and at the end of the entire study) at the end of the study | 730 days
The risk of drug-resistant epilepsy at any point of the study | 730 days
Occurrence of adverse events within the blinded phase of the study | 730 days
Number of adverse events across the whole study | 730 days
Parameters of physical development (weight gain history) across the whole study | 730 days
Parameters of physical development (height gain history) across the whole study | 730 days

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Kotulska-Jozwiak, Principal Investigator — The Children's Memorial Health Institute
Locations (2):
- Poland (2):
  - Medical University of Warsaw, Department of Pediatric Neurology, Warsaw
  - Children's Memorial Health Institute, Neurology and Epileptology, Warsaw